CLINICAL TRIAL: NCT01581320
Title: A Multicenter, Randomized, Double-blind, Active-controlled, Phase III Clinical Trial to Evaluate the Efficacy and Safety of DP-R206 and Bonviva for the Improvement of Vitamin D in Postmenopausal Women With Osteoporosis
Brief Title: Phase III Clinical Trial of DP-R206 and Bonvia In Postmenopausal Women With Osteoporosis
Acronym: DIOS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alvogen Korea (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DP-CTR206-03
Record Dates: First submitted 2012-02-26; First posted 2012-04-20 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2012-04

CONDITIONS: Postmenopausal Women With Osteoporosis
MeSH Terms: interventions — DP-R206; Drug Evaluation; Ibandronic Acid; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- DP-R206 (Experimental)
  Interventions: Drug: Test group
- Bonviva (Active Comparator)
  Interventions: Drug: Reference group

INTERVENTIONS:
Drug: Test group — Once a month, administration of DP-R206 & placebo for 16 weeks
  Other Names: DP-R206 (Test drug); <Ibandronate 150mg + cholecalciferol(Vitamin D3) 24,000IU>
  Arms: DP-R206
Drug: Reference group — Once a month, administration of Bonviva & placebo for 16 weeks
  Other Names: Bonviva®; (Ibandronate 150mg)
  Arms: Bonviva

SUMMARY:
A multicenter, randomized, double-blind, active-controlled, phase III clinical trial to evaluate the efficacy and safety of Dp-R206 and Bonviva for 16 weeks once a month on the improvement of vitamin D in postmenopausal women with osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

* Female more than 40 years old in postmenopausal

Exclusion Criteria:

* Subject who has a history of malignant cancer

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2011-12; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
A ratio of subject whose 25 OHD concentration is less than 15ng/mL | 16weeks
  A ratio of subject whose 25 OHD concentration is less than 15ng/mL after 16weeks

SECONDARY OUTCOMES:
A ratio of subject whose 25 OHD concentration is less than 9ng/mL | 16 weeks
  A ratio of subject whose 25 OHD concentration is less than 9ng/mL after 16weeks
Safety evaluation (AE, Lab test, Vital sign etc) | 16weeks

CONTACTS AND LOCATIONS:
Overall Officials: Moo-il Kang, MD, PhD, Study Chair — The Catholic University of Korea
Locations (1):
- The Catholic University of Korea Seoul St. Mary's Hospital, Seoul, South Korea